CLINICAL TRIAL: NCT00612729
Title: Influence of Light-filters in IOLs on Color Perception and Contrast Acuity. A Randomized, Double-masked Study With Intraindividual Comparison.
Brief Title: Light Filters in Intraocular Lenses (IOLs) and Its Influence on Colour and Contrast Vision.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Hietzing (Other)
Responsible Party: Matthias Wirtitsch MD, Dept. of Ophthalmology, Hospital Hietzing, Vienna, Austria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ye-Or 2008
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2008-12

CONDITIONS: Cataract
Keywords: intraocular lens; light filtering intraocular lens; contrast acuity; color vision
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Polylens Y30 intraocular lens — cataract surgery
Procedure: Orange Series Model PC 440 Y intraocular lens — cataract surgery

SUMMARY:
Visible-light-filtering IOLs are implanted increasingly often in cataract surgery. Several studies examined the effect of light-filters on contrast and colour vision. However, the study outcomes were varying. The present study investigated the effect of two light-filtering IOL on colour perception and contrast acuity using highly sensitive measurement methods.

DETAILED DESCRIPTION:
Prospective, randomized, double-masked study with intraindividual comparison. Implantation of a Polylens Y30 IOL in one eye and an Orange Series Model PC 440 Y in the contralateral eye.

ELIGIBILITY:
Inclusion Criteria:

* bilateral age-related cataract
* age 55 to 80 years
* expected postoperative visual acuity of at least 1.0

Exclusion Criteria:

* amblyopia
* corneal scars
* diabetes
* arterial hypertonia
* pseudoexfoliation-syndrome
* earlier ocular surgeries or laser treatments
* intraocular tumors
* color abnormalities
* expected postoperative visual acuity lower 1.0

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
contrast acuity | 3 month after surgery

SECONDARY OUTCOMES:
visual acuity and color vision | 3 month after surgery
colour perception | 3 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matthias G Wirtitsch, MD, Principal Investigator — Dept of Ophthalmology, Hietzing Hospital, Vienna, Austria; Nadja Karnik, MD, Study Chair — Dept of Ophthalmology, Hietzing Hospital, Vienna, Austria
Locations (1):
- Department of Ophthalmology, Hietzing Hospital, Vienna, Austria